CLINICAL TRIAL: NCT01361438
Title: A Multicenter Total Therapy Strategy for De Novo Adult Philadelphia Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia (ALL) Patients. GIMEMA Protocol LAL1509, EudraCT Number 2010-019119-39
Brief Title: De Novo Adult Philadelphia Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia (ALL) Patients
Acronym: LAL1509
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1509
Record Dates: First submitted 2011-05-13; First posted 2011-05-26 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: ALL Ph Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Total therapy approach — Total therapy approach

SUMMARY:
This study will enroll adult de novo Ph+ acute lymphoblastic leukemia (ALL) patients (≥18 years, ≤60 years). Induction treatment will consist of 12 weeks of Dasatinib oral administration (140 mg QD). Patients will initiate treatment with steroids 7 days prior to starting Dasatinib and will continue up to day 31. Patients will continue treatment with Dasatinib up to day 84, except for disease progression, intolerable toxicity, or withdrawal from study.

DETAILED DESCRIPTION:
This study will enroll adult de novo Ph+ acute lymphoblastic leukemia (ALL) patients (≥18 years, ≤60 years). Induction treatment will consist of 12 weeks of Dasatinib oral administration (140 mg QD). Patients will initiate treatment with steroids 7 days prior to starting Dasatinib and will continue up to day 31. Patients will continue treatment with Dasatinib up to day 84, except for disease progression, intolerable toxicity, or withdrawal from study.

Thereafter:

* patients in hematological and molecular CR will receive a post-remissional treatment consisting of Dasatinib alone for a 6 months period
* patients in hematological CR with persistence of molecular disease will be allografted or, if not eligible or a donor is not available, treated with 2 cycles of a Clofarabine-Cyclophosphamide schedule.

After allograft:

* MRD negative patients (i.e. in CHR and PCR negative) will receive a 6 months Dasatinib maintenance treatment;
* MRD positive patients (i.e. in CHR and PCR positive) will receive Dasatinib as maintenance treatment until relapse or progression.

Patients not transplanted and treated with Clofarabine/Cyclophosphamide will also receive Dasatinib as maintenance treatment until relapse or progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo Ph+ and/or BCR/ABL+ ALL.
* Age ≥18 years old ≤60 years.
* No prior treatment with any anti-leukemic drugs with the exception of steroids for no more than 14 days (including the 7-day pretreatment already scheduled in the protocol).
* WHO performance status ≤2.
* No evidence of central nervous system (CNS) leukemia.
* Normal serum level of potassium, total calcium corrected for serum albumin magnesium and phosphorus, or correctable with supplements.
* ALT and AST ≤2.5 x ULN or ≤5.0 x ULN if considered due to leukemia.
* Alkaline phosphatase ≤2.5 x ULN unless considered to leukemia.
* Serum bilirubin ≤2 x ULN.
* Serum creatinine ≤3 x ULN.
* Serum amylase ≤1.5 x ULN and serum lipase ≤1.5 x ULN.
* Normal cardiac function.
* Written informed consent prior to any study procedures being performed. In addition, patients must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent.

Exclusion Criteria:

* Impaired cardiac function, including any one of the following:

  * LVEF <45% as determined by MUGA scan or echocardiogram.
  * Complete left bundle branch block.
  * Use of a cardiac pacemaker.
  * ST depression of >1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads.
  * Congenital long QT syndrome.
  * History of or presence of significant ventricular or atrial arrhythmia.
  * Clinically significant resting bradycardia (<50 beats per minute).
  * QTc >450 msec on screening ECG (using the QTcF formula).
  * Right bundle branch block plus left anterior hemiblock, bifascicular block.
  * Myocardial infarction within 3 months prior to starting Dasatinib.
  * Angina pectoris.
  * Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Dasatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Use of therapeutic warfarin.
* Acute or chronic liver or renal disease considered unrelated to leukemia.
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Active uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GMCSF) ≤1 week prior to starting study drug.
* Patients who are currently receiving treatment with any of the medications listed in "Appendix H" and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug. The medications listed in "Appendix H" have the potential to prolong the QT interval.
* Patients who have received any antileukemic agents and treatments including steroids. for more than 14 days including 7 days pretreatment that is part of the protocol.
* Patients who have received any investigational drug in the last 2 weeks.
* Patients who have undergone major surgery ≤2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who are pregnant or adults of reproductive potential not employing an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of Dasatinib. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory).
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Non compliant to oral medication patients.
* Significant pleural effusion on baseline chest X-Ray (CXR) or pericardial effusion on baseline echocardiogram.
* Use of H2 blockers or proton pump inhibitors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the trial is to estimate the feasibility of a total therapy strategy in de novo adult Ph positive ALL. | at 42 months
  The primary endpoint is the rate of patients alive in CHR who have completed the trial treatment according to the therapeutic strategy;

SECONDARY OUTCOMES:
The median value of the minimum of PCR levels achieved in each patient during the Dasatinib treatment within day +85, whenever achieved from the start of the Dasatinib. | at 42 months
The rate of patients who become PCR negative after Dasatinib induction. | at 42 months
Out of patients who become PCR negative after induction, the rate of patients who remain persistently negative during maintenance treatment with Dasatinib (without chemotherapy or allogeneic transplant). | at 42 months
The median value of the minimum of PCR levels achieved in each patient after an allogeneic transplant or Clofarabine-Cyclophosphamide treatment as consolidation therapy. | at 42 months
The rate of patients alive in CHR who have completed the maintenance program with Dasatinib after an allogeneic transplant or two cycles of Clofarabine-Cyclophosphamide as consolidation therapy. | at 42 months
Disease free survival estimation starting from the date of evaluation of CHR. | at 42 months
Cumulative incidence of relapse estimation starting from the date of evaluation of CHR. | at 42 months
Overall survival estimation starting from date of inclusion. | at 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foà, Pr., Study Chair — Università Sapienza di Roma
Locations (51):
- Italy (51):
  - Centro Oncologico Basilicata, Rionero in Vulture, Potenza
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - Dipartimento Area Medica P.O., Ascoli Piceno
  - Az. Ospedaliera S. G. Moscati, Avellino
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna
  - Osp. Reg. A. Di Summa, Brindisi
  - CTMO - Ematologia - Ospedale "Binaghi", Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Clinica Ematologica - Università degli Studi, Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - ASL Le1 P.O. Vito Fazzi - U.O. di Ematologia, Lecce
  - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte" di Messina, Messina
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Ospedale Niguarda " Ca Granda", Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Servizio Sanitario Nazionale - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" - Struttura Complessa di Ematologia - Div. TERE, Napoli
  - Prof. D'Arco, Nocera Inferiore
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga, Orbassano
  - Ospedale Cervello, Palermo
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - Div. di Ematologia IRCCS Policlinico S. Matteo, Pavia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Università di Pisa Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Div. di Ematologia, Pisa
  - Ematologia - Ospedale San Carlo, Potenza
  - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Umberto I di Roma - Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Policlinico di Tor Vergata, Rome
  - Ospedale S.Eugenio, Rome
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari
  - Struttura Complessa Ematologia - Azienda Sanitaria Locale BAT1- Presidio Ospedaliero Bisceglie-Trani, Trani
  - U.O. di Ematologia - Azienda Ospedaliera - Pia Fondazione di Culto e di Religione Card. G.Panico, Tricase
  - Policlinico Universitario - Clinica Ematologia, Udine
  - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it